CLINICAL TRIAL: NCT04309981
Title: Pilot Study of the Infusion of Differentiated Autologous T-cells From Peripheral Blood, Expanded and Transduced With a Lentivirus to Express a Chimeric Antigen Receptor With Anti-BCMA (TNFRSF17) Specificity Humanized Conjugated With the Co-stimulatory Region 4-1BB and Signal-transduction CD3z (ARI0002h) in Patients With Relapsed/Refractory Multiple Myeloma With Previous Treatment With Proteasome Inhibitor, Immunomodulatory Drug and Anti-CD38 Monoclonal Antibody
Brief Title: Clinical Trial Using Humanized CART Directed Against BCMA (ARI0002h) in Patients With Relapsed/Refractory Multiple Myeloma to Proteasome Inhibitors, Immunomodulators and Anti-CD38 Antibody.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sara V. Latorre (Other)
Collaborators: Fondos ARI (Assistencia Recerca Intensiva) (Unknown); Instituto de Salud Carlos III (Other Government); Fondo Social La Caixa (Unknown)
Responsible Party: Sponsor-Investigator, Sara V. Latorre, Clinical Research Manager, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTBCMA-HCB-01; 2019-001472-11 (EudraCT Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARI0002h (Experimental): Adult differentiated autologous T-cells from peripheral blood, expanded and transducted with a lentivirus to express a chimeric antigen receptor with anti-BCMA (TNFRSF17) specificity conjugated to the 4-1BB co-stimulatory region and signal-transduction CD3z that has been humanized
  Interventions: Biological: Adult differentiated autologous T-cells with anti-BCMA specificity

INTERVENTIONS:
Biological: Adult differentiated autologous T-cells with anti-BCMA specificity — After pretreatment, adult differentiated autologous T-cells with a chimeric antigen receptor with anti-BCMA specificity will be transfused.
  Other Names: CARTBCMA

SUMMARY:
To assess the safety and efficacy of CARTBCMA ARI0002h in patients with relapsed/refractory multiple myeloma who have received treatment with proteasome inhibitor, immunomodulatory drug and anti-CD38 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18 and 75 years with diagnosis of multiple myeloma
* Disease measurable by monoclonal component in serum and/or urine or by free light chains in serum according to the eligibility criteria for clinical trials of the International Myeloma Working Group
* Previous two or more lines of treatment. Patients must have received at least a proteasome inhibitor (such as bortezomib or carfilzomib), an immunomodulatory drug (lenalidomide or pomalidomide) and an anti-CD38 monoclonal antibody (such as daratumumab)
* Refractory to the last line of treatment
* ECOG functional status ranging from 0 to 2
* Life expectancy over 3 months
* Patients who, after being informed, give their consent by signing the Informed Consent document.

Exclusion Criteria:

* Previous allogeneic transplant in the prior 6 months to inclusion or GVHD that requires active systemic immunosuppressive treatment
* Absolute lymphocyte count <0.1x10^9/ L
* Previous neoplasia, except if patients have been in complete remission > 3 years, except for cutaneous carcinoma (non-melanoma)
* Active infection that requires treatment
* Active infection by HIV, HBV or HCV.
* Uncontrolled medical disease
* Severe organic condition that meets any of the following criteria: EF <40%, DLCO <40%, EGFR <50 ml / min, bilirubin> 3 times normal value (except Gilbert syndrome)
* Previous diagnosis of symptomatic AL amyloidosis
* Pregnant or lactating women. Women of childbearing age should have a negative pregnancy test in the screening phase
* Women of childbearing age, including those whose last menstrual cycle was in the year prior to screening, who cannot or do not wish to use highly effective contraceptive methods from the beginning until the end of the study.
* Men who cannot or do not wish to use highly effective contraceptive methods from the beginning to the end of the study.
* Contraindication to receive conditioning chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 months
Cytokine release syndrome rate | within 30 days of first infusion

SECONDARY OUTCOMES:
Duration of the response | up to 36 months after treatment
Response rate | over the first year
Complete response rate (CR) | at month 3 and month 6 of first infusion
Overall response rate (ORR) | at month 6 of first infusion
Time to complete response | up to 36 months after treatment
Response rate of extramedullary disease by PET-CT | up to 36 months after treatment
Negative MRD rate in bone marrow | at month 3 and month 6 of first infusion
Response rate of extramedullary disease by PET-TC | at month 3
Progression free survival (PFS) | at month 12, and up to 36 months after treatment
Overall survival (OS) defined as the time elapsed between the infusion of ARI0002h and the death of the patient from any cause | up to 36 months after treatment
Presence of tumor lysis syndrome | up to 36 months after treatment
Presence of cytokine release syndrome | up to 36 months after treatment
Presence of neurological toxicity | up to 36 months after treatment
Presence of prolonged cytopenia | up to 36 months after treatment
Persistence of CART BCMA ARI0002 in peripheral blood | month 1, 2, 3, 4, 5, 6 and every 6 months until 2 years of follow up
Expression of BCMA | at screening, at day +28, at day +100, at month 6, 12, 18 and 24
Levels of soluble BCMA in serum | at screening, at day 0, +3, +7,+14,+28, +70 +100, at month 4, 5, 6, 7, 8, 9, 1,11, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernandez de Larrea, MD,PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (7):
- Spain (7):
  - Hospital U. de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zugasti I, Tormo-Ratera M, Oliver-Caldes A, Soler-Perromat JC, Gonzalez-Calle V, Moreno DF, Cabanas V, Lopez-Munoz N, Bartolome-Solanas A, Espanol-Rego M, Reguera-Ortega JL, Rosinol L, Lopez-Corral L, Tovar N, Rodriguez-Lobato LG, Alvarez Perez RM, Varea S, Olesti E, Gomez-Grande A, Frutos L, Tamayo P, Juan M, Moraleda JM, Urbano-Ispizua A, Gonzalez-Navarro EA, Martinez-Lopez J, Mateos MV, Tomas X, Setoain X, Fernandez de Larrea C. Clinical impact of [18F]FDG-PET/CT in ARI0002h treatment, a CAR-T against BCMA for relapsed/refractory multiple myeloma. Blood Adv. 2025 Feb 11;9(3):571-582. doi: 10.1182/bloodadvances.2024014360. PMID 39602341
- [Derived] Oliver-Caldes A, Gonzalez-Calle V, Cabanas V, Espanol-Rego M, Rodriguez-Otero P, Reguera JL, Lopez-Corral L, Martin-Antonio B, Zabaleta A, Inoges S, Varea S, Rosinol L, Lopez-Diaz de Cerio A, Tovar N, Jimenez R, Lopez-Parra M, Rodriguez-Lobato LG, Sanchez-Salinas A, Olesti E, Calvo-Orteu M, Delgado J, Perez-Simon JA, Paiva B, Prosper F, Saez-Penataro J, Juan M, Moraleda JM, Mateos MV, Pascal M, Urbano-Ispizua A, Fernandez de Larrea C. Fractionated initial infusion and booster dose of ARI0002h, a humanised, BCMA-directed CAR T-cell therapy, for patients with relapsed or refractory multiple myeloma (CARTBCMA-HCB-01): a single-arm, multicentre, academic pilot study. Lancet Oncol. 2023 Aug;24(8):913-924. doi: 10.1016/S1470-2045(23)00222-X. Epub 2023 Jul 3. PMID 37414060
- [Derived] Oliver-Caldes A, Jimenez R, Espanol-Rego M, Cibeira MT, Ortiz-Maldonado V, Quintana LF, Castillo P, Guijarro F, Tovar N, Montoro M, Benitez-Ribas D, Bataller A, Gonzalez-Navarro EA, Cid J, Lozano M, Perez-Amill L, Martin-Antonio B, Mena MP, Moreno DF, Rodriguez-Lobato LG, Campistol JM, Calvo G, Blade J, Rosinol L, Juan M, Pascal M, Urbano-Ispizua A, Fernandez de Larrea C. First report of CART treatment in AL amyloidosis and relapsed/refractory multiple myeloma. J Immunother Cancer. 2021 Dec;9(12):e003783. doi: 10.1136/jitc-2021-003783. PMID 34876408